CLINICAL TRIAL: NCT01955798
Title: Direct Trocar Entry Versus Veress Needle Entry in Laparoscopic Gynecological Surgery , a Randomized Study
Brief Title: Direct Trocar Entry Versus Veress Needle Entry in Laparoscopic Gynecological Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IP Change Hospital
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Ignacio Rodriguez MSc, Epidemilolgy, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX2013001
Record Dates: First submitted 2013-09-20; First posted 2013-10-08 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Laparoscopic Gynecological Surgery
Keywords: Laparoscopy; Gyneacological; Entry techniques
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trocar (Experimental): Pyramidal tip reusable 11mm trocar
  Interventions: Procedure: Laparoscopic direct entry Trocar; Device: Trocar
- Veress needle (Active Comparator): Veress needle
  Interventions: Procedure: Laparoscopic entry Veress needle; Device: Veress needle

INTERVENTIONS:
Procedure: Laparoscopic direct entry Trocar — Laparoscopic direct entry with trocar
  Arms: Trocar
Procedure: Laparoscopic entry Veress needle — Laparoscopic entry with Veress needle
  Arms: Veress needle
Device: Trocar
  Arms: Trocar
Device: Veress needle
  Arms: Veress needle

SUMMARY:
The Veress needle is the laparoscopic entry technique most commonly used among gynecologists. Direct trocar entry is another method to gain entry to the abdomen that is uncommon to gynecologists.

This prospective and randomized study will compare the two entry techniques with regard to:

* Complications related to the entry technique and previous surgeries
* Time taken to enter the abdomen
* The number of attempts taken to enter the abdomen

DETAILED DESCRIPTION:
Patients of Dexeus Universitary Institute that are having a laparoscopic surgery for gynecological purposes will participate in the study. Patients with previous middle laparotomies or 3 or more abdominal suregeries will be excluded from the study. A patient information sheet will be provided and written consent will be obtained. Patients who give written consent will be randomized into the two arms of the trial. All patient information will be confidential and only be available to researches involved in the study.

Only three expert surgeons of the Gynecological Department of Dexeus Universitary Institute will participate in the study.

300 women will be recruited over a two year period and the data will be analysed by a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Any woman suitable for laparoscopic gyneacological surgery

Exclusion Criteria:

* Previus supra-infra umbilical laparotomy
* three or more previous abdominal surgeries

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Complications during entry in laparoscopy | During surgery
  Complications during entry in laparoscopy like vascular injury, bowel injury,conversion to laparotomy, omental injury, etc

SECONDARY OUTCOMES:
Time to enter in the abdominal cavity | During surgery
  Time in seconds from the impact of the trocar or the veress needle to enter in the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Vazquez, MD, Principal Investigator — Salut de la Mujer Dexeus
Locations (1):
- Hospital Quiron Dexeus, Barcelona, Spain

REFERENCES:
- [Background] Ahmad G, O'Flynn H, Duffy JM, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD006583. doi: 10.1002/14651858.CD006583.pub3. PMID 22336819
- [Background] Tinelli A, Malvasi A, Guido M, Tsin DA, Hudelist G, Stark M, Mettler L. Laparoscopy entry in patients with previous abdominal and pelvic surgery. Surg Innov. 2011 Sep;18(3):201-5. doi: 10.1177/1553350610393989. Epub 2011 Jan 18. PMID 21245070
- See also: Related Info — http://www.dexeus.com